CLINICAL TRIAL: NCT01223807
Title: Effects of a Short-term Diaphragmatic Breathing Training Program in COPD Patients: a Randomized Controlled Trial
Brief Title: Effects of a Diaphragmatic Breathing Training Program in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Wellington Pereira dos Santos Yamaguti, University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: uspferd
Record Dates: First submitted 2010-10-15; First posted 2010-10-19 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2008-06

CONDITIONS: COPD
Keywords: COPD, diaphragm, rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (No Intervention): The control group will receive only usual care.
- Diaphragmatic breathing training (Experimental): The training group will be submitted to a diaphragmatic breathing training program of 4 weeks.
  Interventions: Other: Diaphragmatic breathing training

INTERVENTIONS:
Other: Diaphragmatic breathing training — The training group will participate in a diaphragmatic breathing program which will consist of three 45-min sessions each week (12 sessions totally). The program training will be individualized and supervised by the same physiotherapist. In each session, the patients will be initially instructed to perform 3 series of 10 maximally inspirations, predominantly with abdominal motion, while reducing upper rib cage motion in a supine position.
  Arms: Diaphragmatic breathing training

SUMMARY:
Diaphragmatic dysfunction and alterations of thoracoabdominal motions are common in patients with chronic obstructive pulmonary disease (COPD). Several studies have described an impairment in diaphragmatic mobility of COPD patients compared to age matched control subjects and it has been associated with increase in dyspnea, exercise intolerance and mortality. COPD patients also experiment a higher activity of the accessory breathing muscles, which greatly increases the work of breathing and dyspnea sensation.

Breathing strategies have been considered an important component of pulmonary rehabilitation and refer to a range of techniques, including/which includes the diaphragmatic breathing (DB). The principal aim of DB is to improve the participation of the abdominal motion while reducing the accessory muscles activity. The role of DB as an adjunctive treatment modality in the rehabilitation of COPD patients remains controversial. Despite the conflicting results, improvement of the abdominal motion and a reduction of thoracic excursion, during voluntarily DB, has been described as a common finding of several studies. The investigators hypothesized that a 4-week DBTP could induce higher participation of the diaphragm and this modification would relieve respiratory symptoms and improve exercise tolerance and the HRQoL. Therefore, in this randomized controlled trial the investigators aimed to test the effects of a short-term DBTP on thoracoabdominal motion, pulmonary function, diaphragmatic mobility, dyspnea, HRQoL and exercise tolerance in patients with mild to severe COPD.

ELIGIBILITY:
Inclusion Criteria: (1) age between 50 and 80 years; (2) a post-bronchodilator forced expiratory volume in one second (FEV1) < 80% of the predicted value and a FEV1/ forced vital capacity (CVF) ratio < 0,7; (3) stable respiratory/clinical condition without changes in medication and symptoms (dyspnea, volume or color of sputum) for at least 4 weeks before admission to the study; and (4) receiving regular treatment with inhaled bronchodilators and steroids.

Exclusion Criteria: (1) presence of other pulmonary, cardiovascular or musculoskeletal diseases; (2) previously participation in any exercise-training program in the last 2 years before participating in this study; and (3) current smokers.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-06; Primary Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
thoracoabdominal motion | 2 years

SECONDARY OUTCOMES:
diaphragmatic mobility | 2 years

REFERENCES:
- [Derived] Yamaguti WP, Claudino RC, Neto AP, Chammas MC, Gomes AC, Salge JM, Moriya HT, Cukier A, Carvalho CR. Diaphragmatic breathing training program improves abdominal motion during natural breathing in patients with chronic obstructive pulmonary disease: a randomized controlled trial. Arch Phys Med Rehabil. 2012 Apr;93(4):571-7. doi: 10.1016/j.apmr.2011.11.026. PMID 22464088